# A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Parallel-group Study to Assess the Safety and Efficacy of ASP4345 as Add-on Treatment for Cognitive Impairment in Subjects with Schizophrenia on Stable Doses of Antipsychotic Medication

ISN/Protocol 4345-CL-0015

ClinicalTrials.gov Identifier: NCT03557931

Date of Statistical Analysis Plan: 22 Aug 2019

**Sponsor:** Astellas Pharma Global Development, Inc. (APGD)

1 Astellas Way Northbrook, IL 60062

# STATISTICAL ANALYSIS PLAN

Final Version 2.0 dated 22-August-2019

A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Parallel-group Study to Assess the Safety and Efficacy of ASP4345 as Add-on Treatment for Cognitive Impairment in Subjects with Schizophrenia on Stable Doses of Antipsychotic Medication

ISN: 4345-CL-0015

Astellas Pharma Global Development, Inc. (APGD)

This document contains confidential information which is the intellectual property of Astellas. By accepting or reviewing this document, you agree to hold this information in confidence and not copy or disclose it to others or use it for unauthorized purposes except (1) as otherwise agreed to in writing; (2) where required by applicable law; (3) where disclosure is directly related to the care and safety of the research participant; and (4) where disclosure of such information is made to a member of the investigator's team who agrees to hold this information in confidence.

# **Table of Contents**

| I. | | LIS | T OF ABBREVIATIONS AND KEY TERMS······ 4 |
|---|---|---|---|
| 1 | | INT | TRODUCTION 7 |
| 2 | | STU | JDY OBJECTIVE(S) AND DESIGN···································· |
| | 2.1 | | Study Objective(s) · · · · · 7 |
| | | 2.1.1 | Primary Objectives ······ 7 |
| | | 2.1.2 | Secondary Objectives · |
| | | 2.1.3 | Exploratory Objectives |
| | 2.2 | 2 | Study Design 8 |
| | 2.3 | 3 | Randomization 8 |
| 3 | | SAI | MPLE SIZE9 |
| 4 | | AN | ALYSIS SETS ·····9 |
| | 4.1 | l | Full Analysis Set ···· 9 |
| | | 4.1.1 | Modified Full Analysis Set 1 ····· 9 |
| | | 4.1.2 | Modified Full Analysis Set 2 ····· 9 |
| | 4.2 | 2 | Intent-to-Treat Set |
| | 4.3 | 3 | Safety Analysis Set ······10 |
| | 4.4 | | Pharmacokinetics Analysis Set ·······10 |
| 5 | | EFI | FICACY ENDPOINTS ······10 |
| | 5.1 | l | Primary Efficacy Endpoint(s) |
| | 5.2 | 2 | Secondary Efficacy Endpoints · |
| | 5.3 | | Exploratory Efficacy Endpoints · · · · · · 10 |
| 6 | | STA | ATISTICAL METHODOLOGY ······11 |
| | 6.1 | | General Considerations |
| | 6.2 | 2 | Study Population |
| | | 6.2.1 | Disposition of Subjects · · · · · 11 |
| | | 6.2.2 | Protocol Deviations · · · · · · 12 |
| | | 6.2.3 | Demographic and Other Baseline Characteristics · · · · · · 12 |
| | | 6.2.4 | Previous and Concomitant Medications · · · · · 12 |
| | 6.3 | 3 | Study Drugs Exposure and Compliance 12 |
| | 6.4 | 1 | Analysis of Efficacy · · · · · · 13 |
| | | 6.4.1 | Analysis of Primary Efficacy Endpoint(s)······13 |

| | 6.4.2 | | Analysis of Secondary Efficacy Endpoints15 |
|---|---|---|---|
| | | | Analysis of Exploratory Endpoints · · · · · · 16 |
| | 6.5 | | Analysis of Safety 18 |
| | 6.: | | Adverse Events · · · · · 18 |
| | 6.5.2 | | Clinical Laboratory Evaluation · · · · · 19 |
| | | 6.5.3 | Vital Signs·····20 |
| | | 6.5.4 | Electrocardiograms ······21 |
| | | 6.5.5 | Metabolic Parameters21 |
| | | 6.5.6 | Columbia-Suicide Severity Rating Scale ······21 |
| | | 6.5.7 | Movement Disorder (Abnormal Involuntary Movement Scale) ······21 |
| | | 6.5.8 | Simpson Angus Scale ———————————————————————————————————— |
| | | 6.5.9 | Barnes Akathisia Rating Scale · · · · · 22 |
| | 6.6 | 5 | Analysis of Pharmacokinetic ———————————————————————————————————— |
| | | 6.6.1 | Estimation of Pharmacokinetic Parameters ······22 |
| | 6.7 | | Interim Analysis (and Early Discontinuation of the Clinical Study)22 |
| | 6.7 | / | interin Analysis (and Early Discontinuation of the Clinical Study) |
| | 6.8 | | Additional Conventions23 |
| | | | Additional Conventions |
| | | 6.8.1<br>6.8.2 | Additional Conventions |
| 7 | | 6.8.1<br>6.8.2 | Additional Conventions |
| 7 | | 6.8.1<br>6.8.2<br><b>REV</b> | Additional Conventions |
| | | 6.8.1<br>6.8.2<br><b>REV</b> | Additional Conventions 23 Analysis Windows 23 Imputation Rules for Incomplete Dates 25 VISION AND RATIONALE 26 |
| 8 | | 6.8.1<br>6.8.2<br>REV | Additional Conventions |
| 8 | 6.8 | 6.8.1<br>6.8.2<br><b>REV</b><br><b>API</b> | Additional Conventions 23 Analysis Windows 23 Imputation Rules for Incomplete Dates 25 VISION AND RATIONALE 26 ERENCES 26 PENDICES 27 Appendix 1: Author and Approver Signatures 27 Appendix 2: Adverse Events of Special Interest (Preferred Terms; MedDRA |
| 8 | 9.1 | 6.8.1<br>6.8.2<br><b>REV</b><br><b>API</b> | Additional Conventions 23 Analysis Windows 23 Imputation Rules for Incomplete Dates 25 VISION AND RATIONALE 26 FERENCES 26 PENDICES 27 Appendix 1: Author and Approver Signatures 27 |
| 8 | 9.1 | 6.8.1<br>6.8.2<br><b>REV</b><br><b>API</b> | Additional Conventions 23 Analysis Windows 23 Imputation Rules for Incomplete Dates 25 VISION AND RATIONALE 26 ERENCES 26 PENDICES 27 Appendix 1: Author and Approver Signatures 27 Appendix 2: Adverse Events of Special Interest (Preferred Terms; MedDRA |
| 8 | 9.1 | 6.8.1<br>6.8.2<br>REV<br>API | Additional Conventions 23 Analysis Windows 23 Imputation Rules for Incomplete Dates 25 VISION AND RATIONALE 26 FERENCES 26 PENDICES 27 Appendix 1: Author and Approver Signatures 27 Appendix 2: Adverse Events of Special Interest (Preferred Terms; MedDRA 18.0) 28 |

# I. LIST OF ABBREVIATIONS AND KEY TERMS

#### List of Abbreviations

| List of Abbreviations | |
|---|---|
| Abbreviations | Description of abbreviations |
| AE | adverse event |
| AIMS | Abnormal Involuntary Movement Scale |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| ANCOVA | Analysis of Covariance |
| APGD | Astellas Pharma Global Development, Inc. |
| ASSR | auditory steady-state response |
| AST | aspartate aminotransferase |
| AUC | area under the concentration-time curve |
| BARS | Barnes Akathisia Rating Scale |
| BMI | body mass index |
| CGI-S | Clinical Global Impression of Severity Scale |
| CI | confidence interval |
| CIAS | cognitive impairment associated with schizophrenia |
| C <sub>max</sub> | maximum concentration |
| COMT | catechol-o-methyltransferase |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| CV | coefficient of variation |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| ЕоТ | end-of-treatment |
| ET | early termination |
| FAS | full analysis set |
| HDL | high-density lipoprotein |
| IRT | Interactive Response Technology |
| LDH | lactate dehydrogenase |
| LDL | Low-density lipoprotein |
| LS | least squares |
| MATRICS | Measurement and Treatment Research to Improve Cognition in Schizophrenia |
| MATRICS-CT | Measurement and Treatment Research to Improve Cognition in Schizophrenia |
| | Coprimary and Translations |
| MCCB | Measurement and Treatment Research to Improve Cognition in Schizophrenia<br>Consensus Cognitive Battery |
| MedDRA | medical dictionary for regulatory activities |
| MMRM | Mixed Models Repeated Measures |
| NSA-16 | Negative Symptom Assessment Scale |
| NSAIDs | non-steroidal anti-inflammatory drugs |
| PANSS | Positive and Negative Symptom Scale |
| <u></u> | <u> </u> |

**Sponsor:** Astellas Pharma Global Development, Inc. (APGD) ISN/Protocol 4345-CL-0015

| Abbreviations | Description of abbreviations |
|---|---|
| PGx | pharmacogenetic |
| PKAS | pharmacokinetic analysis set |
| QD | daily |
| QTcF | QT interval using Fridericia's formula |
| SAE | serious adverse event |
| SAF | safety analysis set |
| SAP | statistical analysis plan |
| SAS | Simpson Angus Scale |
| SE | standard error |
| TEAE | treatment emergent adverse events |
| TSH | thyroid-stimulating hormone |
| ULN | upper limit of normal |
| UPSA-2-ER | University of California San Diego Performance-based Skills Assessment-2 |
| | Extended Range |

**Sponsor:** Astellas Pharma Global Development, Inc. (APGD) ISN/Protocol 4345-CL-0015

# **List of Key Terms**

| Terms | Definition of terms |
|---|---|
| Baseline | The last measurement/evaluation on or prior to the first dose of randomized |
| | therapy is considered the baseline measure/evaluation. |
| Endpoint | Variable that pertains to the efficacy or safety evaluations of a trial. |
| Enroll | To register or enter a subject into a clinical trial. NOTE: Once a subject has |
| | received the study drug or placebo, the clinical trial protocol applies to the subject. |
| Intervention | The drug, device, therapy or process under investigation in a clinical study that |
| | is believed to have an effect on outcomes of interest in a study. (e.g., health-related quality of life, efficacy, safety, pharmacoeconomics). |
| Investigational | Period of time where major interests of protocol objectives are observed, and |
| period | where the test drug or comparative drug (sometimes without randomization) is |
| | usually given to a subject, and continues until the last assessment after |
| | completing administration of the test drug or comparative drug. |
| Post investigational | Period of time after the last assessment of the protocol. Follow-up |
| period | observations for sustained adverse events and/or survival are done in this |
| | period. |
| Randomization | The process of assigning trial subjects to treatment or control groups using an |
| ranaomization | element of chance to determine assignments in order to reduce bias. |
| Screening | A process of active consideration of potential subjects for enrollment in a trial. |
| Screen failure | Potential subject who did not meet 1 or more criteria required for participation in a trial. |
| Screening period | Period of time before entering the investigational period, usually from the time |
| | when a subject signs the consent until just before the test drug or comparative |
| | drug (sometimes without randomization) is given to a subject. |
| Study period | Period of time from the first site initiation date to the last site completing the |
| | study. |
| Variable | Any entity that varies; any attribute, phenomenon or event that can have |
| | different qualitative or quantitative values. |

#### 1 INTRODUCTION

This Statistical Analysis Plan (SAP) contains technical and detailed elaboration of the principal features of the analysis described in the protocol, and includes procedures for executing the statistical analysis to fulfil the objectives of the study.

SAP Final Version 2.0

The final SAP will be approved prior to database hardlock and unblinding the subject treatment assignment.

Critical changes that affected the statistical analyses from the analyses planned in the SAP will be documented in the Clinical Study Report (CSR).

## 2 STUDY OBJECTIVE(S) AND DESIGN

## 2.1 Study Objective(s)

The objectives of the study, conducted in subjects with cognitive impairment associated with schizophrenia, are the following:

#### 2.1.1 Primary Objectives

- To evaluate the efficacy of ASP4345 on cognitive impairment compared to placebo using change from baseline in MATRICS Consensus Cognitive Battery (MCCB) neurocognitive composite score (excluding social cognition domain). The primary estimand will use a Hypothetical Strategy and compare patients as though they had continued on the assigned treatment.
- To evaluate the safety and tolerability of ASP4345 compared to placebo

#### 2.1.2 Secondary Objectives

- To evaluate the effects of ASP4345 compared to placebo on functional capacity using the University of California San Diego Performance-based Skills Assessment-2 Extended Range (UPSA-2-ER) total score.
- To evaluate the pharmacokinetic profile of ASP4345 and its metabolites, if necessary

#### 2.1.3 Exploratory Objectives

- To evaluate the effects of ASP4345 compared to placebo using:
  - o the 16-item version of the Negative Symptom Assessment Scale (NSA-16)
  - o the individual domains of the MCCB
  - o the assessment of general clinical symptoms with the Positive and Negative Symptom Scale (PANSS)
  - o the assessment of the Clinical Global Impression of Severity Scale (CGI-S)
- To evaluate the relationship between the CGI-S and MCCB neurocognitive composite score
- To evaluate the relationship between number of cognitive training levels, including repeat levels, completed (as a measure of compliance with cognitive training) and MCCB neurocognitive composite score
- To evaluate the pharmacogenetic impact on ASP4345 pharmacodynamic results

# 2.2 Study Design

This is a randomized, double-blind, placebo-controlled, 3-arm oral dose study to evaluate the safety and efficacy of ASP4345 in subjects with cognitive impairment associated with schizophrenia on stable doses of risperidone, quetiapine, olanzapine, ziprasidone, aripiprazole, brexpiprazole, paliperidone or lurasidone for at least 4 weeks prior to screening for oral medications and 2 months for depot medications. The study will consist of the following periods:

- Screening period (up to 28 days)
- Double-blind treatment period (12 weeks/84 days)
- Follow-up period (14 days post last dose)

Approximately 420 subjects are planned to be screened with up to 210 subjects enrolled in 1 of 3 arms. Study groups will consist of approximately 90 placebo subjects and 60 subjects each per active study arm randomized in 3:2:2 ratio to receive 1 of 2 doses of ASP4345 or matching placebo daily (QD) for 12 weeks. Study treatment assignments will be according to the following table:

| Group | Dose Regimen | Number |
|-------|--------------|--------|
| A | 50 mg, QD | 60 |
| В | 150 mg, QD | 60 |
| C | Placebo, QD | 90 |

All subjects will be administered the first dose of blinded study drug at the site following randomization and provided with mobile applications that provide supplemental cognitive training and record treatment compliance. Subjects will return to the clinic weekly for safety, efficacy, and/or pharmacokinetic procedures at days 7, 14, 21, 28, 35, 42, 49, 56, 63, 70, 77 and 84. Subjects will continue their antipsychotic treatment for the entire study and will be followed for 14 days after their last dose of study drug.

Subjects terminating early from the study treatment will be encouraged to complete scheduled visits. All subjects are allowed to stop study drug, but continue in the study through day 84 according to the current visit schedule unless the participant specifically withdraws consent for any further contact with him/her or persons previously authorized by the participant provide this information.

#### 2.3 Randomization

Subjects will be randomized in a 3:2:2 ratio to a treatment arm (placebo to active) according to the randomization schedules through IRT. All subjects who meet the eligibility criteria will be randomized. The site personal will dispense the treatment according to the IRT system's assignment. Randomization will occur by site (stratified by site). In order to reduce the impact of incomplete blocks at any given site, a Latin square design will be used to generate the randomization list such that blocks are balanced both in regard to the number of treatment assignments but also to the order in which treatments are assigned. Blocks will be

dynamically assigned by the IRT system to sites once they request a randomization number, so that all blocks in a Latin square will be assigned before moving on to the next Latin square.

#### 3 SAMPLE SIZE

A total sample size of 210 subjects will be randomized in 3:2:2 ratio (approximately 90 placebo and 60 subjects each per active study arm) into 1 of 2 doses of ASP4345 or matching placebo. The sample size will provide approximately 82% power for the pairwise comparisons to placebo to detect an effect size of at least 0.43 in the primary outcome measure, assuming a 1 sided 5% significance level, with statistical significance achieved at an effect size of approximately 0.28. Note that the decision criteria to proceed with the development of the compound will be based on effect sizes rather than statistical significance. The number of subjects planned for this clinical study are considered sufficient to achieve the clinical study objectives.

#### 4 ANALYSIS SETS

In accordance with International Conference on Harmonization (ICH) recommendations in guidelines E3 and E9, the following analysis sets will be used for the analyses.

The determination of whether subjects are included or excluded from the safety and efficacy analysis sets will be made prior to database hard-lock. All classifications can be made programmatically and so a Classificiation meeting may not be held.

# 4.1 Full Analysis Set

The full analysis set (FAS) will consist of all subjects who are randomized and receive at least one dose of study drug and have at least one post baseline MCCB measurement. This will be the primary analysis set for efficacy analyses.

#### 4.1.1 Modified Full Analysis Set 1

A modified full analysis set 1 (mFAS1) will be a subset of the FAS, with the exclusion of subjects whose study coordinator may have become unblinded during the study due to an error in the drug accountability system, and where the subejet's rater is the same person as the study coordinator.

#### 4.1.2 Modified Full Analysis Set 2

A modified full analysis set 2 (mFAS2) will be a subset of the FAS, with the exclusion of subjects whose study coordinator may have become unblinded during the study due to an error in the drug accountability system.

#### 4.2 Intent-to-Treat Set

The Intent-to-Treat analysis set (ITT) will consist of all subjects who are randomized into the study. The ITT will be used to assess the robustness of the results of the primary efficacy endpoint from the statistical tests based on the FAS. Select demographic and baseline characteristics may also be summarized for the ITT.

#### 4.3 Safety Analysis Set

The Safety Analysis Set (SAF) consists of all subjects who took at least 1 dose of study drug, and will be used for safety analyses.

For the statistical summary of the safety data, the SAF will be used.

## 4.4 Pharmacokinetics Analysis Set

The pharmacokinetic analysis set (PKAS) consists of all subjects who took at least 1 dose of study drug and who have at least 1 plasma concentration.

The PKAS will be used for all summaries and analyses of the pharmacokinetic data.

#### 5 EFFICACY ENDPOINTS

# 5.1 Primary Efficacy Endpoint(s)

- Change from baseline to week 12/EoT for ASP4345 compared to placebo for the MCCB neurocognitive composite score (excluding social cognition domain).
- Safety and Tolerability:
  - o Nature, frequency and severity of AEs.
  - Vital signs (sitting or supine blood pressure, pulse and body temperature)
  - Clinical laboratory tests (hematology, biochemistry [including cystatin C, serum prolactin, and ACTH] and urinalysis)
  - o Routine 12-lead ECG
  - o Columbia-Suicide Severity Rating Scale (C-SSRS)
  - Changes in individual indices of metabolic syndrome (weight, waist circumference, cholesterol, triglycerides, high-density lipoprotein [HDL; the second screening visit and day 77), and hemoglobin A1c [HbA1c]
  - Movement disorder (Abnormal Involuntary Movement Scale [AIMS], Simpson Angus Scale [SAS] and Barnes Akathisia Rating Scale [BARS])

# 5.2 Secondary Efficacy Endpoints

- Change from baseline to week 12/EoT for ASP4345 compared to placebo for the UPSA 2 ER instrument total score
- Pharmacokinetics:
  - o ASP4345 and its metabolites, if necessary (plasma): C<sub>trough</sub>.

# 5.3 Exploratory Efficacy Endpoints

- Change from baseline to week 12/EoT for ASP4345 compared to placebo for the NSA-16 only for the subjects who have at least 1 negative symptom of at least moderate severity
- Change from baseline to week 12/EoT for ASP4345 compared to placebo for the MCCB composite score.
- Change from baseline to week 12/EoT for ASP4345 compared to placebo for each of the MCCB domains.
- Change from baseline to week 12/EoT for ASP4345 compared to placebo for the PANSS
- Change from baseline to week 12/EoT for ASP4345 compared to placebo for the CGI-S

Sponsor: Astellas Pharma Global Development, Inc. (APGD) SAP Final Version 2.0

ISN/Protocol 4345-CL-0015

• Correlation between MCCB and CGI-S scores at each measurement (weeks -4, -3, 0, 6, 12)

- Correlation between change from baseline to week 12/EoT in MCCB and change from baseline to week 12/EoT in CGI-S scores
- Correlation between the number of cognitive training levels, including repeat levels, completed (as a measure of compliance with cognitive training) and MCCB neurocognitive composite score
- Pharmacogenetics:
  - Catechol-o-methyltransferase (COMT) and dopamine D<sub>1</sub> and D<sub>3</sub> receptor genotyping

#### 6 STATISTICAL METHODOLOGY

#### 6.1 General Considerations

Continuous data will be summarized descriptively including the number of subjects (n), mean, standard deviation (SD), median, minimum and maximum. Categorical data will be summarized by frequencies and percentages. Percentages by categories will be based on the number of subjects with no missing data, i.e. the percentages for the non-missing categories will add up to 100%.

A 2-sided significance level of 0.10, unless otherwise specified, will be used for all statistical tests on efficacy endpoints without multiplicity adjustment.

All data summarization and analyses will be performed using SAS® Version 9.3 or higher on Unix. Specifications for table, figures, and data listing formats can be found in the TLF specifications.

# 6.2 Study Population

Analysis of the primary efficacy endpoint will be conducted on the FAS and ITT. The interpretation of results from statistical tests will be based on the FAS. The ITT will be used to assess the robustness of the results from the statistical tests based on the FAS. Analysis of the secondary and exploratory efficacy endpoints will be done on the FAS only.

Data such as patient disposition, demographics and baseline characteristics will be summarized for FAS in the event that the definition of FAS is identical to SAF (i.e., if no patients were given wrong study drug and all have a post-baseline MCCB neurocognitive composite score). If FAS is not identical to SAF then data will be summarized for both FAS and SAF as specified in the relevant sections.

#### 6.2.1 Disposition of Subjects

Disposition of subjects will be summarized for the FAS by treatment group and overall. Number of subjects who complete or prematurely discontinue from the treatment or study (ie, follow up period) will be summarized by treatment group and overall. For the discontinuation, the primary reason reported by the investigator will be summarized.

Number and percentage of subjects for each analysis set will be summarized by treatment group and overall.

#### **6.2.2** Protocol Deviations

The number and percentage of subjects with the following protocol deviation criteria will be summarized for each criterion and overall, by treatment group and total as well as by investigative site. Subjects deviating from a criterion more than once will be counted once for the corresponding criterion.

The unique identifiers will be as follows:

- PD1 Entered into the study even though they did not satisfy entry criteria,
- PD2 Developed withdrawal criteria during the study and was not withdrawn,
- PD3 Received wrong treatment or incorrect dose,
- PD4 Received excluded concomitant treatment.

#### 6.2.3 Demographic and Other Baseline Characteristics

Demographic, age, sex, race, ethnicity, weight, height, BMI, and smoking status, and other baseline characteristics will be summarized descriptively by treatment group and overall for the FAS, ITT and SAF.

Medical history is coded in MedDRA, and will be summarized by System Organ Class (SOC) and Preferred Term (PT), by treatment group and overall for the SAF.

Medical and psychiatric history for each subject will be presented in a listing.

#### 6.2.4 Previous and Concomitant Medications

Previous and concomitant medications will be summarized by therapeutic subgroup (ATC 2nd level) and chemical subgroup (ATC 4th level) and preferred WHO name by treatment group for the FAS. Subjects taking the same medication multiple times will be counted once per medication and investigational period. A medication which can be classified into several chemical and/or therapeutic subgroups is presented in all chemical and therapeutic subgroups.

Medications taken for treatment of schizophrenia during the 12 months prior to screening and other medication taken 28 days prior to the screening visit and up to the first dose of study medication (treatment period) will be defined as prior schizophrenia medications or other prior medication, respectively. Concomitant medications are defined as any medications that patients took after the first dose of study medication and through last dose of study drug. Medications that started prior to first administration of study drug and continued while study drug was given will be counted in both previous and concomitant medications.

# **6.3** Study Drugs Exposure and Compliance

Duration and compliance of study drug will be summarized for FAS, ITT, and SAF by treatment group and overall.

Number and percentages of subjects with the following categories of study drug duration will be summarized: >0 to  $\le 2$  days, >2 to  $\le 7$  days, >7 to  $\le 14$  days, >14 to  $\le 21$  days, >21 to  $\le 42$  days, >42 to  $\le 56$  days, >56 to  $\le 84$  days.

Number and percentages of subjects with the following cumulative categories of study drug duration will be summarized:  $\geq 1$  days,  $\geq 7$  days,  $\geq 14$  days,  $\geq 28$  days,  $\geq 28$  days,  $\geq 42$  days, and  $\geq 56$  days.

Study drug compliance will be summarized and listed both for product accountability from an IRT system as well as from daily virtual monitoring by use of a mobile application. Product accountability will be the primary source of compliance, and % compliance will be calculated at each visit and overall as ([the number of pills dispensed] – [the number of pills returned]) / [the number of pills expected consumed] \* 100, where the number of pills expected consumed is the duration in days.

# 6.4 Analysis of Efficacy

## 6.4.1 Analysis of Primary Efficacy Endpoint(s)

No multiplicity adjustment will be necessary in this study.

#### 6.4.1.1 Primary Analysis for Primary Efficacy Endpoint(s)

Consistent with the Hypothetical Strategy used for the estimand which is to compare patients as though they had continued on the assigned treatment, MMRM will use all available ontreatment data to inform end of treatment mean treatment effect estimates without requiring explicit imputation for missing data (i.e., for discontinued subjects). There will be no adjustment made for multiple comparisons. The primary analysis will use the FAS.

The MCCB neurocognitive composite score is a standardized mean of the six domain scores (excluding social cognition). Raw scores are converted to age and sex adjusted t-scores which are standardized to normative data, and have a mean of 50 and standard deviation of 10 in the general healthy population. A higher score indicates less impairment.

The primary endpoint of change from baseline in MCCB neurocognitive composite T score will be analyzed using a Mixed Models Repeated Measures (MMRM) approach. The model will contain fixed effect terms for treatment group, pooled site, visit (the repeated term), treatment by visit, and visit by baseline, with the MCCB neurocognitive composite score at baseline used as a covariate. Pooled centers will be generated and documented prior to database lock. If the inclusion of pooled centers creates modeling problems, then dropping that factor will be considered. Subject will be identified as subject in the repeated statement. Residuals from the model will be tested for normality using the Shapiro-Wilk test; if the normality assumption is rejected then data transformations will be explored. If necessary, the model may be run on ranked values as a non-parametric alternative. An unstructrured covariance structure will be used initially, if the model fails to converge other covariance structures will be explored. The Kenward-Roger method of estimation of degrees of freedom and the restricted maximum likelihood (REML) method will be used.

Least squares (LS) means (± standard error [SE]) and 2-sided 90% CIs and p-values for the LS mean treatment differences between each dose of ASP4345 and placebo will be presented for the primary endpoint. Effect size (Cohen's d) will also be shown, as:

**Sponsor:** Astellas Pharma Global Development, Inc. (APGD)

ISN/Protocol 4345-CL-0015

$$d_s = t\sqrt{\frac{1}{n_1} + \frac{1}{n_2}}$$

where t is the t-value for the least squares mean pairwise difference of ASP4345 vs placebo from the MMRM model.

There will be two hypotheses tested. Hypothesis 1 is given as follows:

 $H_{0A}$ : The LS mean change from baseline at week 12 for Group A (50 mg ASP4345) and Group C (placebo) are the same

H<sub>1A</sub>: The LS mean change from baseline at week 12 for Group A (50 mg ASP4345) and Group C (placebo) are not the same

Hypothesis 2 is given as follows:

 $H_{0B}$ : The LS mean change from baseline at week 12 for Group B (150 mg ASP4345) and Group C (placebo) are the same

 $H_{1B}$ : The LS mean change from baseline at week 12 for Group B (150 mg ASP4345) and Group C (placebo) are not the same

#### 6.4.1.2 Sensitivity Analysis for Primary Efficacy Endpoint(s)

The relationship between the number of cognitive training levels, including repeat levels completed at week 12, (as a measure of compliance with cognitive training) and MCCB neurocognitive composite end of treatment scores will be evaluated using correlations overall and by treatment group.

Additionally, the primary efficacy analysis as defined in section 6.4.1.1 will be conducted using mFAS1 and mFAS2.

#### 6.4.1.2.1 Cognitive Training

The number of training levels completed as well as the percentage of the number expected completed will be summarized. The percent of the number of training levels completed out of the number expected completed will be calculated as: [number of levels played / expected number of levels] \* 100, where the expected number of training levels will increase in a step fashion, by 48 on day 1, day 7, day 14 and so on (as shown in the table below). In between 'steps', i.e. from day 1 until day 7, regardless of whether a subject completes the entire week the expected number of training levels will be constant. Additionally, training task performance will be assessed prior to the start of cognitive training (pre assessment) and again after the last cognitive training (post assessment) with a standardized task assessment (Sound Sweeps) to evaluate improvement. Pre, post and change pre to post values will be summarized.

**Sponsor:** Astellas Pharma Global Development, Inc. (APGD)

ISN/Protocol 4345-CL-0015

| Week | Interval | Increase in Expected | Cumulative Expected Number of |
|------|----------------|----------------------|-------------------------------|
| | | Number of Training | Training Levels |
| | | Levels at Start of | |
| | | Interval | |
| 1 | Day 1 to <7 | 48 | 48 |
| 2 | Day 7 to <14 | 48 | 96 |
| 3 | Day 14 to <21 | 48 | 144 |
| 4 | Day 21 to <28 | 48 | 192 |
| 5 | Day 28 to <35 | 48 | 240 |
| 6 | Day 35 to <42 | 48 | 288 |
| 7 | Day 42 to <49 | 48 | 336 |
| 8 | Day 49 to <56 | 48 | 384 |
| 9 | Day 56 to <63 | 48 | 432 |
| 10 | Day 63 to <70 | 48 | 480 |
| 11 | Day 70 to <77 | 48 | 528 |
| 12 | Day 77 to <=84 | 48 | 576 |

An additional interval may be added for subjects with extended treatment periods. Incomplete intervals will be normalized to the expected interval.

#### 6.4.1.3 Subgroup Analysis for Primary Efficacy Endpoint(s)

The primary outcome of neurocognitive MCCB score will be summarized by subgroups. The subgroups (categories) will be:

- Duration of diagnosis (>10 years,  $\leq$  10 years)
- Type of diagnosis (schizophrenia, schizoaffective)
- Smoking status (current, non-smoker ([including former])
- Sex (male, female)
- Cannabis use (3 groups based on laboratory results: Never positive, positive pre-dose or week 12, positive predose and week 12; where positive pre-dose is positive week 0 and/or screening)
- Compliance based on electronic mobile application (<85% compliance, ≥85% compliance)

#### 6.4.2 Analysis of Secondary Efficacy Endpoints

The secondary efficacy endpoint of change from baseline to week 12/EoT in the UPSA-2 Extended Range instrument will be analyzed using ANCOVA, in each of the six domains and a total score. The model will contain terms for treatment group and pooled site, with the corresponding score at baseline used as a covariate.

LS means (± SE) and 2-sided 90% CIs for the LS mean treatment differences between each dose of ASP4345 and placebo will be presented as for the primary endpoint. There will be no adjustment made for multiple comparisons.

The sensitivity analysis described in 6.4.1.2 and the subgroups described in section 6.4.1.3 will also be completed for the secondary efficacy endpoint.

SAP Final Version 2.0

#### 6.4.3 Analysis of Exploratory Endpoints

Exploratory endpoints listed below will be analyzed using the same MMRM model as the primary efficacy analysis.

- Change from baseline to week 12/EoT for NSA-16 total negative score, only for the subjects who have at least 1 negative symptom of moderate severity at baseline (a score ≥3 or ≤6 for one of the 16 symptoms assessed)
- Change from baseline to week 12/EoT for NSA-16 global negative symptoms rating
- Change from baseline to week 12/EoT for the MCCB composite T score
- Change from baseline to week 12/EoT for each of the seven MCCB domain T scores
- Change from baseline to week 12/EoT for the PANSS total score
- Change from baseline to week 12/EoT for ASP4345 compared to placebo for the CGI-S
- The pharmacogenetics test listed below will be measured at baseline only. Genotyping data will be analyzed and reported separatelyfrom the rest of the study data.
  - Catechol-o-methyltransferase (COMT) and dopamine D<sub>1</sub> and D<sub>3</sub> receptor genotyping

The NSA-16 consists of 16 negative symptoms with scores of 0-6 for each item. Scores of 9 (not able to rate) will not be included in any continuous summary statistics. Scores for five factors (Communication, Emotion/Affect, Social Involvement, Motivation and Retardation) will be calculated. If all item have scores  $\geq 0$  and  $\leq 6$ , each factor score is the sum of all the items in that factor. If there are missing items (including ratings of 9) within a factor, provided the number missing is  $\leq 34\%$  the factor score will be calculated as the sum of all items within the factor, with the missing item imputed as the average score of the observed items.

A factor score will not be calculated if the number missing is greater than 34%, and if any factor score is not calculated the total score will be not be calculated. Provided all factor scores are calculated, the total negative score will be the sum of all factor scores..

- Communication [4 items; minimum number of items to calculate factor score is 3]
  - o Q1, Prolonged time to respond
  - o Q2, Restricted speech quantity
  - o Q3, Impoverished speech content
  - o Q4, Inarticulate speech
- Emotion/Affect [3 items; minimum number of items to calculate factor score is 2]
  - o Q5, Reduced range
  - o Q6, Reduced modulation of intensity
  - o Q7, Reduced display on demand
- Social Involvement [3 items; minimum number of items to calculate factor score is 2]
  - o O8, Reduced social drive
  - Q9, Poor rapport with interviewer

**Sponsor:** Astellas Pharma Global Development, Inc. (APGD) ISN/Protocol 4345-CL-0015

- o Q10, Interest in Emotional and Physical Intimacy
- Motivation [4 items; minimum number of items to calculate factor score is 3]
  - o Q11, Poor grooming and hygiene
  - o Q12, Reduced sense of purpose
  - o Q13, Reduced interests
  - o Q14, Reduced daily activity
- Retardation [2 items; minimum number of items to calculate factor score is 2]
  - o Q15, Reduced expressive gestures
  - O Q16, Slowed movements

A higher score indicates more severe symptoms. A global negative symptoms rating (a scale ranging from '1=No evidence of negative symptoms' to '7=Extremely severe negative symptoms (incapacitating)' is also assessed.

For patients who have at least one negative symptom of at least moderate severity (a score  $\geq 3$  or  $\leq 6$  for one of the 16 symptom assessments), the negative symptom burden will be further assessed with the total negative score, as calculated above. Continuous descriptive statistics for each factor score, the total negative symptom score and the global negative symptoms rating will be shown, along with the number and percentage in each category for the individual 16 symptom scores, by treatment and week.

PANSS total score is the summation of ratings across all 30 items. Traditional PANSS subscores are calculated as follows:

- Positive score: summation of ratings across 7 positive items (P1 to P7)
- Negative score: summation of ratings across 7 negative items (N1 to N7)
- General psychopathology score: summation of ratings across 16 general psychopathology items (G1 to G16).
- Composite score: positive score negative score

In addition, five factors are calculated as follows:

- Anergia: summation of N1, N2, G7 and G10
- Thought Disturbance: summation of P2, P3, P5 and G9
- Activation: summation of P4, G4 and G5
- Paranoid / Belligerence: summation of P6, P7 and G8
- Depression: summation of G1, G2, G3 and G6

PANSS total score, sub-scores, five factors and associated changes from baseline will be listed and summarized by treatment and visit. The PANSS individual item ratings will be listed.

The Clinical Global Impression of Severity Scale (CGI-S) is a 7-point scale rating the severity of a patient's illness. Continuous descriptive statistics as well as the number and percentage in each category will be shown by treatment and week. The relationship between MCCB and CGI-S will be examined as follows:

**Sponsor:** Astellas Pharma Global Development, Inc. (APGD) SAP Final Version 2.0

ISN/Protocol 4345-CL-0015

• Correlation between MCCB and CGI-S scores at each measurement (weeks -4, -3, 0, 6, 12)

• Correlation between change from baseline to week 12/EoT in MCCB and change from baseline to week 12/EoT in CGI-S scores

## 6.5 Analysis of Safety

#### **6.5.1** Adverse Events

AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). Treatment Emergent Adverse Event (TEAE) is defined as an AE observed after starting administration of the study drug and 28 days after the last dose of study drug. A study drug-related TEAE is defined as any TEAE with at least possible relationship to study treatment as assessed by the investigator or with missing assessment of the causal relationship. There are two types of adverse events of special interest: TEAEs related to abuse, and TAEAs related to drug withdrawal. See appendix 2 for a complete list of the MedDRA preferred AE terms to be included in each AE of special interest type.

An overview table will include the following:

- Number of TEAEs
- Number and percentage of subjects with TEAEs
- Number of drug related TEAEs
- Number and percentage of subjects with causally drug related TEAEs
- Number of serious TEAEs
- Number and percentage of subjects with serious TEAEs
- Number of serious drug related TEAEs
- Number and percentage of subjects with serious drug related TEAEs
- Number of TEAEs leading to withdrawal of treatment
- Number and percentage of subjects with TEAEs leading to withdrawal of treatment, and
- Number of deaths
- Number of TEAEs leading to death
- Number and percentage of subjects with TEAEs leading to death
- Number of drug related TEAEs leading to death
- Number and percentage of subjects with drug related TEAEs leading to death
- Number of TEAEs of special interest related to abuse during the treatment period
- Number of TEAEs of special interest related to abuse during the follow up period
- Number of TEAEs of special interest related to drug withdrawal during the treatment period
- Number of TEAEs of special interest related to drug withdrawal during the follow up period

The number and percentage of subjects with TEAEs, as classified by SOC, and PT will be summarized for each treatment group. Summaries will be provided for the following:

- TEAEs
- drug related TEAEs

Sponsor: Astellas Pharma Global Development, Inc. (APGD) SAP Final Version 2.0

ISN/Protocol 4345-CL-0015

- drug related TEAEs by severity
- drug related TEAEs leading to death
- serious TEAEs
- drug related serious TEAEs
- TEAEs by severity
- TEAEs leading to death
- TEAEs leading to withdrawal of treatment
- drug related TEAEs leading to withdrawal of treatment
- Common (>=5% in Any Treatment Group) TEAEs excluding serious adverse events
- TEAEs of special interest related to abuse during the treatment period
- TEAEs of special interest related to abuse during the follow up period
- TEAEs of special interest related to drug withdrawal during the treatment period
- TEAEs of special interest related to drug withdrawal during the follow up period

The number of TEAEs and the number and percentage of subjects with TEAEs, as classified by SOC and PT will be summarized by severity and by relationship to study drug. In the subject count, if a subject has multiple TEAEs with the same SOC or PT, but with differing severity or relationship, then the subject will be counted once with the worst severity and highest degree of relationship. If any of the severity or relationship values are missing then the subject will be counted only once with missing severity or relationship.

The number and percentage of subjects with TEAEs, as classified by SOC and PT will be summarized for each treatment group by time interval. For each adverse event in a particular interval, a subject will be counted if there is an onset of a treatment-emergent adverse event regardless of onset in other intervals.

Time intervals will be categorized according to the following categories:

- less than 7 days
- o at least 7 days, less than 14 days
- o at least 14 days, less than 28 days
- o at least 28 days, less than 42 days
- 42 days or more

Following data will be presented graphically by treatment group:

- Overview of TEAEs using dot-and-forest plot
- TEAEs by SOC using dot-and-forest plot

#### 6.5.2 Clinical Laboratory Evaluation

The baseline value will be the last non-missing value taken on or prior to day of first dose of study drug. Quantitative values evaluated by the central laboratory including hematology, biochemistry, and urinalysis will be summarized using mean, standard deviation, minimum, maximum and median by treatment group at each analysis visit. Additionally, a within-subject change will be calculated as the post-baseline measurement minus the baseline measurement and summarized in the same way. Each laboratory result will be classified as low (L), normal (N), or high (H) at each visit according to the laboratory supplied reference

ranges. The number and percentage of subjects below and above reference range will be summarized for each treatment group at each visit.

For hematology and biochemistry, a summary of shifts of reference range changes from baseline to worst finding during the treatment period will be presented for each treatment group.

The following data will be presented graphically by treatment group:

Change from baseline in laboratory test results using box plot

#### 6.5.2.1 Liver Safety Assessment

The liver safety assessments will be summarized by the following categories below based on the measurements from Alkaline Phosphatase (ALP), Alanine Transaminase (ALT), total bilirubin, Aspartate Transaminase (AST) and their combination are defined. These parameters will be measured from a central laboratory.

The subject's highest value during the investigational period (day of first dose and through 1 day of the last dose of study drug) will be used.

- ALT > 3xULN, > 5xULN, > 10xULN, > 20xULN
- AST > 3xULN, > 5xULN, > 10xULN, > 20xULN
- ALT or AST > 3xULN, > 5xULN, > 10xULN, > 20xULN
- ALP > 1.5xULN
- Total Bilirubin >2xULN
- (ALT or AST > 3xULN) and Total Bilirubin > 2xULN
- (ALT or AST > 3xULN) and ALP< 2xULN and Total Bilirubin > 2xULN

The last 2 criteria where 2 or more parameters are evaluated will be with the measurements on the same day or up to a maximum of 1 day apart.

The denominator for each criterion will be the number of subjects who have at least one value during the investigational period. The number and percentage of subjects meeting the criteria during the investigational period will be summarized by treatment group.

#### 6.5.3 Vital Signs

The baseline value will be the last non-missing value taken on or prior to day of first dose of study drug.

Vital signs (systolic blood pressure, diastolic blood pressure, and pulse rate) will be summarized by treatment group and visit. Additionally, a within-subject change will be calculated at each visit as the post-baseline measurement minus the baseline measurement and summarized by treatment group and visit. Analysis visits are defined in the Analysis Windows section 6.8.1

#### 6.5.4 Electrocardiograms

ECG variables will be summarized using mean, standard deviation, minimum, maximum and median for each treatment group at each treatment visit and time point, including changes from baseline.

Number and percent of subjects with normal, not clinically significant abnormal, and clinically significant abnormal results as assessed by investigator for the 12 lead ECG will be tabulated by treatment group at each treatment visit and time point.

The QTcF interval will be summarized using frequency tables for each treatment visit and time point for values of clinical importance using the range criteria below.

| | QTcF Interval Criteria Value (msec) |
|------------------------|--------------------------------------|
| Normal | $\leq$ 450 males; $\leq$ 470 females |
| Borderline | > 450 males; > 470 females |
| Prolonged | > 480 males; > 490 females |
| Clinically significant | > 500 males; > 500 females |

The QTcF interval will also be summarized by the frequencies of subjects with a change from baseline of clinical importance using the criteria identified below. These summaries will be provided for each treatment visit and time point.

| Variable | Change from Baseline |
|----------------------|----------------------|
| QTcF Interval (msec) | > 30 |
| | > 60 |

Differences between treatments in the frequency of changes greater than 30, and greater than 60, will be evaluated with the Chi-square test at each treatment visit.

#### 6.5.5 Metabolic Parameters

Descriptive statistics will be used to summarize individual indices of metabolic syndrome results (weight, waist circumference, cholesterol, triglycerides, HDL [the second screening visit and day 77], and fasting glucose), and hemoglobin A1c [HbA1c] and changes from baseline by treatment group and time point. Differences between treatments in change from baseline will be assessed with same MMRM model as the primary efficacy analysis, with the exception of HDL which will be analyzed using the same ANCOVA model as the secondary analysis.

## 6.5.6 Columbia-Suicide Severity Rating Scale

Number and percentage of subjects in each of the categories of C-SSRS, as well as changes from baseline, will be summarized by treatment group and visit.

#### 6.5.7 Movement Disorder (Abnormal Involuntary Movement Scale)

Number and percentage of subjects in each rating category will be summarized for each of the items of the AIMS by treatment group and visit. A total score will be calculated as the sum of items 1 through 7 and descriptive statistics will be used to summarize the total score

at each visit as well as changes from baseline. Differences between treatments in the total score will be evaluated with the same MMRM model as the primary efficacy analysis.

#### 6.5.8 Simpson Angus Scale

Number and percentage of subjects in each rating category will be summarized for each of the items of the SAS by treatment group and visit. Total scores will be calculated as the sum of each item, and categorized as [<3 (normal); 3-5 (minimal); 6-11 (clinically significant); 12-17 (severe); ≥18 (extreme)]. Descriptive statistics will be used to summarize the total score (sum) and total score (categorical) at each visit as well as changes from baseline. Differences between treatments in categorical total scores will be evaluated with a general estimating equations (GEE) model. The model will contain terms for treatment group, pooled site, visit (the repeated term), and treatment by visit, with the categorical score at baseline used as a covariate. Odds ratios comparing each active treatment and control will be assessed at week 6 and week 12.

## 6.5.9 Barnes Akathisia Rating Scale

Number and percentage of subjects in each of the categories of BARS will be summarized by treatment group and visit. Differences between treatments in the Global Clinical Assessment of Akathisia, scored from 0 (absent) to 5 (severe akathisia), will be evaluated with a general estimating equations (GEE) model. The model will contain terms for treatment group, pooled site, visit (the repeated term), and treatment by visit, with the Global Clinical Assessment of Akathisia score at baseline used as a covariate. Odds ratios comparing each active treatment and control will be assessed at week 6 and week 12.

# 6.6 Analysis of Pharmacokinetic

Descriptive statistics (e.g., N, mean, standard deviation, minimum, median, maximum, coefficient of variation [CV], geometric mean, and geometric CV) will be provided for plasma concentrations of ASP4345 and possible metabolite(s) by time point.

#### 6.6.1 Estimation of Pharmacokinetic Parameters

Population pharmacokinetic model will be developed based on ASP4345 plasma concentration data obtained from subjects who have at least 1 pharmacokinetic sample. Population pharmacokinetics and/or pharmacokinetic/pharmacodynamics analyses will be performed by modeling and simulation scientist. All details of the population pharmacokinetic analysis will be described in a separate analysis plan and a separate population pharmacokinetic modeling report will be written.

# 6.7 Interim Analysis (and Early Discontinuation of the Clinical Study)

There will be no interim analysis.

# 6.8 Additional Conventions

# 6.8.1 Analysis Windows

The data summary by visits will be done following the analysis windows specified in the tables below:

# MCCB, NSA-16, ECG, Weight & Waist, Global Impression of Severity Scale, AIMS, BARS, and SAS Analysis Windows:

| <b>Analysis Visits</b> | Scheduled Day in Protocol | Analysis Windows (day) |
|---|---|---|
| Baseline (Week 0) | Day 1 | Last non-missing value between -28 and 1 |
| | | (inclusive) |
| Week 6 | Day 42 | 35 to 49 |
| Week 12 | Day 84 | 77 to 91 |
| Week 12/ET | Day 84 | ≥ 2 |

#### **UPSA-2-ER Analysis Windows:**

| <b>Analysis Visits</b> | Scheduled Day in Protocol | Analysis Windows (day) |
|---|---|---|
| Baseline (Week 0) | Day 1 | Last non-missing value between -28 and 1 |
| | | (inclusive) |
| Week 12 | Day 84 | 77 to 91 |
| Week 12/ET | Day 84 | ≥ 2 |

#### **Vital Signs Analysis Windows:**

| Analysis Visits | Scheduled Day in Protocol | Analysis Windows (day) |
|---|---|---|
| Baseline (Week 0) | Day 1 | Last non-missing value between -28 and 1 |
| | | (inclusive) |
| Week 1 | Day 7 | 2 to 10 |
| Week 2 | Day 14 | 11 to 17 |
| Week 3 | Day 21 | 18 to 24 |
| Week 4 | Day 28 | 25 to 31 |
| Week 5 | Day 35 | 32 to 38 |
| Week 6 | Day 42 | 39 to 45 |
| Week 7 | Day 49 | 46 to 52 |
| Week 8 | Day 56 | 53 to 59 |
| Week 9 | Day 63 | 60 to 66 |
| Week 10 | Day 70 | 67 to 73 |
| Week 11 | Day 77 | 74 to 80 |
| Week 12 | Day 84 | 81 to 112 |
| Week 12/ET | Day 84 | $\geq 2$ |

**Sponsor:** Astellas Pharma Global Development, Inc. (APGD)

ISN/Protocol 4345-CL-0015

# Columbia-Suicide Severity Rating Scale Analysis Windows:

| <b>Analysis Visits</b> | Scheduled Day in Protocol | Analysis Windows (day) |
|---|---|---|
| Baseline (Week 0) | Day 1 | Last non-missing value between -28 and 1 |
| | | (inclusive) |
| Week 1 | Day 7 | 2 to 10 |
| Week 2 | Day 14 | 11 to 17 |
| Week 3 | Day 21 | 18 to 24 |
| Week 4 | Day 28 | 25 to 31 |
| Week 5 | Day 35 | 32 to 38 |
| Week 6 | Day 42 | 39 to 45 |
| Week 7 | Day 49 | 46 to 52 |
| Week 8 | Day 56 | 53 to 59 |
| Week 9 | Day 63 | 60 to 66 |
| Week 10 | Day 70 | 67 to 73 |
| Week 11 | Day 77 | 74 to 80 |
| Week 12 | Day 84 | 81 to 112 |
| Week 12/ET | Day 84 | ≥ 2 |
| Week 14 | Day 98 | 91 to 105 |

# Positive and Negative Symptom Scale Analysis Windows:

| Analysis Visits | <b>Scheduled Day in Protocol</b> | Analysis Windows (day) |
|---|---|---|
| Baseline (Week 0) | Day 1 | Last non-missing value between -28 and 1 |
| | | (inclusive) |
| Week 2 | Day 14 | 7 to 21 |
| Week 6 | Day 42 | 35 to 49 |
| Week 12 | Day 84 | 77 to 91 |
| Week 12/ET | Day 84 | ≥ 2 |

# Laboratory (Hematology, Full Biochemistry, and Urinalysis) Analysis Windows:

| <b>Analysis Visits</b> | Scheduled Day in Protocol | Analysis Windows (day) |
|---|---|---|
| Baseline (Week 0) | Day -1 | Last non-missing value between -28 and 1 |
| | | (inclusive) |
| Week 5 | Day 35 | 28 to 42 |
| Week 11 | Day 77 | 70 to 84 |
| Week 11/ET | Day 77 | $\geq 2$ |
| Week 14 | Day 98 | 91 to 105 |

#### Laboratory (Abbreviated Biochemistry) Analysis Windows:

| Analysis Visits | Scheduled Day in Protocol | Analysis Windows (day) |
|---|---|---|
| Baseline (Week 0) | Day 1 | Last non-missing value between -28 and 1 |
| | | (inclusive) |
| Week 1 | Day 7 | 2 to 10 |
| Week 2 | Day 14 | 11 to 17 |
| Week 3 | Day 21 | 18 to 24 |
| Week 4 | Day 28 | 25 to 35 |
| Week 6 | Day 42 | 36 to 45 |
| Week 7 | Day 49 | 46 to 52 |
| Week 8 | Day 56 | 53 to 59 |
| Week 9 | Day 63 | 60 to 66 |
| Week 10 | Day 70 | 67 to 73 |
| Week 10/ET | Day 70 | $\geq 2$ |

If more than one observation exists within the analysis window, the observation closest to the scheduled visit day will be selected for that visit. If there are two observations that have the same distance from the scheduled day, the value that is after the scheduled day will be selected in the analysis. If more than one observation is made on the same day, an average value if continuous or the worst value if categorical will be included in the analysis.

The Follow Up visit will include all data collected beyond 10 days after the last dose of study drug. If there are more than one value, then the value that is closest to day 28 from the last dose of study drug will be selected for the analysis. The same logic will be applied as in above for more than one value.

#### **6.8.2** Imputation Rules for Incomplete Dates

In case of missing partial start and stop dates for concomitant medications, the following rules will be used:

If the start date is missing or partial:

- if the month is missing, use January
- if the day is missing, use the first day of the month under consideration
- if the year is missing, use year of the informed consent date
- if the entire date is missing, use informed consent date

If the stop date is missing or partial:

- if the month is missing, use December
- if the day is missing, use the last day of the month under consideration
- if the year or the entire date is missing, set the stop date to December 31<sup>st</sup>, 2099

If the imputed start date is after the stop date, then the imputed start date will be 1 day prior to the stop date.

For AEs, a missing or incomplete onset date will be imputed according to the following conventions.

**Sponsor:** Astellas Pharma Global Development, Inc. (APGD)

ISN/Protocol 4345-CL-0015

If an onset date is missing or only the year is known, the imputed onset date will be the date of first dose of study drug.

SAP Final Version 2.0

If only the year is known for the AE onset date, the imputed onset date will be the latest of the following non-missing dates:

- Date of first dose of study drug
- January 1 of the year of AE onset date

If only the month and year is known for the onset date, set the surrogate onset date to the first day of that month and then apply the following rules.

- If the month and year of the onset date is prior to the month and year of the first dose of study drug, then the surrogate onset date will be the imputed onset date.
- If the month and year of the onset date is on or after the month and year of the first dose of study drug, then the imputed onset date will be the <u>latest</u> of the following non-missing dates:
  - Date of first dose of study drug
  - Surrogate onset date

If the imputed onset date is after the adverse event end date, the imputed onset date will be the same as the adverse event end date.

#### 7 REVISION AND RATIONALE

#### 8 REFERENCES

Calulating and reporting effect sizes to facitiltate cumulative science: a practical primer for t-tests and ANOVAs. Lakens, Daniel, *Frontiers in Psychology* November 2013 Vol 4 Article 863.

# 9 APPENDICES

# 9.1 Appendix 1: Author and Approver Signatures

| Prepared by: | | Date: | |
|--------------|-----|-------|--------------------|
| | PPD | | Date (DD Mmm YYYY) |
| Approved by: | | Date: | |
| | PPD | | Date (DD Mmm YYYY) |
| Approved by: | | Date: | |
| | PPD | | Date (DD Mmm YYYY) |

# 9.2 Appendix 2: Adverse Events of Special Interest (Preferred Terms; MedDRA 18.0)

SAP Final Version 2.0

### 9.2.1 Adverse Events of Interest Related to Abuse requiring narratives

**Euphoria-related Terms** 

| Euphoria-related relins | |
|-------------------------|-------------------------|
| Preferred term | Lowest level term |
| Euphoric mood | Feeling high |
| Elevated mood | |
| Feeling abnormal | |
| Feeling drunk | |
| Feeling of relaxation | |
| Thinking abnormal | |
| Hallucination, mixed | |
| Inappropriate affect | |
| | Dizziness and giddiness |

**Dissociative/Psychotic Terms** 

| Preferred term | Lowest level term |
|-----------------|------------------------------|
| Psychosis acute | Psychosis |
| Aggression | |
| | Confusion and disorientation |

Terms Indicative of Impaired Attention, Cognition, Mood, and Psychomotor Events

| Preferred term | Lowest level term |
|---|---|
| Somnolence | |
| Psychomotor hyperactivity/decreased activity | Hyperactivity/hypoactivity |
| | Mood disorders and disturbances |
| | Mental impairment disorders |
| | Drug tolerance, habituation, drug withdrawal |
| | syndrome, substance-related disorders |

**Inappropriate Affect** 

| mappi opi ate i meet | |
|----------------------|------------------------------|
| Preferred term | Lowest level term |
| Inappropriate affect | Elation inappropriate |
| | Exhilaration inappropriate |
| | Inappropriate mood elevation |
| Product tampering | Medication tampering |

# 9.2.2 Drug Abuse – Related Adverse Events

| System Organ<br>Class | Higher Level<br>GT | Higher<br>Level Term | Preferred term | Lower Level Term |
|---|---|---|---|---|
| Psychiatric disorders | Mood | Emotional | Euphoric | Euphoria |
| | disorders and | and mood | Mood | Euphoric |
| | disturbances | disturbances | | Euphoric mood |
| | NEC | NEC | | Exaggerated well- |
| | | | | being |
| | | | | Feeling high |
| | | | | Felt high |
| | | | | High |
| | | | | High feeling |
| | | | | Laughter |
| | | | Mood altered | Affect alteration |
| | | | | Affect altered |
| | | | | Altered mood |
| | | | | Bad mood |
| | | | | Mood alteration |
| | | | | NOS |
| | | | | Mood altered |
| | | | | Mood change |
| | | | Elevated | Elevated mood |
| | | | mood | Mood elevated |
| | | Affect | Inappropriate | Elation |
| | | alterations | affect | inappropriate |
| | | | | Exhilaration |
| | | | | inappropriate |
| | | | | Exhiliration |
| | | | | inappropriate |
| | | | | Feeling happy |
| | | | | inappropriately |
| | | | | Inappropriate affect |
| | | | | Inappropriate crying |
| | | | | Inappropriate |
| | | | | elation |
| | | | | Inappropriate exhilaration |
| | | | | Inappropriate laughter |
| | | | | Inappropriate mood |
| | | | | elevation |
| | | | | Mood elevation |
| | | | | inappropriate |
| | Disturbances | Perception | Hallucination | Drug-induced |
| | in thinking | disturbances | | hallucinosis |

| System Organ | Higher Level | Higher | Preferred | |
|---|---|---|---|---|
| Class | GT | Level Term | term | Lower Level Term |
| | and | | | Hallucinating |
| | perception | | | Hallucination |
| | | | | Hallucination NOS |
| | | | | Hallucinations |
| | | | | Hallucinations |
| | | | | aggravated |
| | | | | Kinesthetic |
| | | | | hallucination |
| | | | | Organic hallucinosis |
| | | | | syndrome |
| | | | | Pseudohallucination |
| | | | | Sensory |
| | | | | hallucinations |
| | | | | Stump hallucination |
| | | | Hallucination, | Auditory |
| | | | auditory | hallucinations |
| | | | | Hallucination |
| | | | | auditory |
| | | | | Hallucination, |
| | | | | auditory |
| | | | | Verbal |
| | | | | hallucinations |
| | | | Hallucination, | Hallucination visual |
| | | | visual | Hallucination with |
| | | | | color |
| | | | | Hallucination with |
| | | | | colour |
| | | | | Hallucination, visual |
| | | | | Visual |
| | | | | hallucinations |
| General disorders | General | Feelings and | Feeling drunk | Drunk-like effect |
| and administration | system | sensations | | Drunkenness feeling |
| site conditions | disorders | NEC | | of The state of |
| | NEC | | D 1: | Feeling drunk |
| | | | Feeling | Cotton wool in head |
| | | | abnormal | Feeling abnormal |
| | | | | Feeling bad |
| | | | | Feeling dazed |
| | | | | Feeling floating |
| | | | | Feeling lifeless |
| | | | | Feeling miserable |
| | | | | Feeling stoned |
| | | | | Feeling strange |

**Sponsor:** Astellas Pharma Global Development, Inc. (APGD) ISN/Protocol 4345-CL-0015

| System Organ<br>Class | Higher Level<br>GT | Higher<br>Level Term | Preferred term | Lower Level Term |
|---|---|---|---|---|
| | | | | Feeling weightless |
| | | | | Feels awful |
| | | | | Feels bad |
| | | | | Feels poorly |
| | | | | Felt like a zombie |
| | | | | Floating feeling |
| | | | | Foggy feeling head |
| | | | | Funny episode |
| | | | | Fuzzy |
| | | | | Fuzzy head |
| | | | | Muzzy head |
| | | | | Neck strange feeling |
| | | | | of |
| | | | | Soft feeling |
| | | | | Spaced out |
| | | | | Thick head |
| | | | | Unstable feeling |
| | | | | Weird feeling |

# 9.2.3 Drug Withdrawal – Related Adverse Events

| | Higher Level GT | Higher Level Term | Preferred Term |
|---|---|---|---|
| Psychiatric disorders | Anxiety disorders | Anxiety symptoms | Agitation |
| | and symptoms | | |
| Nervous system | Neurological | Neurological signs | |
| disorders | disorders NEC | and symptoms NEC | |
| Psychiatric disorders | Depressed mood | Mood alterations | Anhedonia |
| | disorders and | with depressive | |
| | disturbances | symptoms | |
| Psychiatric disorders | Anxiety disorders | Anxiety symptoms | Anxiety |
| | and symptoms | | |
| Musculoskeletal and | Muscle disorders | Muscle related signs | Chills |
| connective tissue | | and symptoms NEC | |
| disorders | | | |
| Musculoskeletal and | Muscle disorders | Feelings and | 1 |
| connective tissue | | sensations NEC | |
| disorders | | | |
| Psychiatric disorders | Depressed mood | Mood alterations | Depressed mood |
| | disorders and | with depressive | |
| | disturbances | symptoms | |
| Psychiatric disorders | Depressed mood | Depressive disorders | Depression |
| J | disorders and | 1 | 1 |
| | disturbances | | |
| Gastrointestinal | Gastrointestinal | Diarrhoea (excl | Diarrhoea |
| disorders | motility and | infective) | |
| | defaecation | , | |
| | conditions | | |
| Psychiatric disorders | Mood disorders and | Emotional and mood | Dysphoria |
| | disturbances | disturbances NEC | |
| Nervous system | Sleep disturbances | Sleep disturbances | Dyssomnia |
| disorders | (incl subtypes) | NEC | |
| Psychiatric disorders | Sleep disorders and | Dyssomnias | 1 |
| | disturbances | | |
| Psychiatric disorders | Depressed mood | Depressive disorders | Dysthymic disorder |
| | disorders and | | |
| | disturbances | | |
| Psychiatric disorders | Depressed mood | Mood alterations | Feeling of despair |
| | disorders and | with depressive | |
| | disturbances | symptoms | |
| Nervous system | Headaches | Headaches NEC | Headache |
| disorders | | | |
| Skin and | Skin appendage | Apocrine and eccrine | Hyperhidrosis |
| subcutaneous tissue | conditions | gland disorders | |
| disorders | | | |
| General disorders | General system | General signs and | |
| and administration | disorders NEC | symptoms NEC | |

| | Higher Level GT | Higher Level Term | Preferred Term |
|---|---|---|---|
| site conditions | | | |
| Psychiatric disorders | Sleep disorders and disturbances | Disturbances in initiating and maintaining sleep | Insomnia |
| Nervous system disorders | Sleep disturbances | Disturbances in initiating and maintaining sleep | |
| Psychiatric disorders | Depressed mood disorders and disturbances | Mood alterations with depressive symptoms | Morose |
| Gastrointestinal disorders | Gastrointestinal signs and symptoms | Nausea and vomiting symptoms | Nausea |
| Psychiatric disorders | Depressed mood disorders and disturbances | Mood alterations with depressive symptoms | Negative thoughts |
| Psychiatric disorders | Anxiety disorders and symptoms | Anxiety symptoms | Nervousness |
| Psychiatric disorders | Anxiety disorders and symptoms | Obsessive-<br>compulsive disorders<br>and symptoms | Obsessive thoughts |
| General disorders<br>and administration<br>site conditions | General system<br>disorders NEC | Pain and discomfort<br>NEC | Pain |
| Nervous system disorders | Sleep disturbances (incl subtypes) | Sleep disturbances<br>NEC | Poor quality sleep |
| Psychiatric disorders | Sleep disorders and disturbances | Dyssomnias | |
| Cardiac disorders | Cardiac disorder signs and symptoms | Cardiac signs and symptoms NEC | Syncope |
| Vascular disorders | Decreased and<br>nonspecific blood<br>pressure disorders<br>and shock | Circulatory collapse and shock | |
| Nervous system disorders | Neurological disorders NEC | Disturbances in consciousness NEC | |
| Psychiatric disorders | Sleep disorders and disturbances | Disturbances in initiating and maintaining sleep | Terminal insomnia<br>(lower level term of<br>interest: early |
| Nervous system disorders | Sleep disturbances | Disturbances in initiating and maintaining sleep | morning awakening) |
| Nervous system disorders | Movement disorders (incl parkinsonism) | Tremor (excl congenital) | Tremor |
| Gastrointestinal disorders | Gastrointestinal signs and symptoms | Nausea and vomiting symptoms | Vomiting |

**Sponsor:** Astellas Pharma Global Development, Inc. (APGD) ISN/Protocol 4345-CL-0015

SAP Final Version 2.0